CLINICAL TRIAL: NCT05636189
Title: Effect of Prewarming During Induction of General Anesthesia Combined With Warmed Intravenous Fluid on Core Temperature in Patients Undergoing Urologic Surgery.
Brief Title: Effect of Prewarming During Induction of General Anesthesia Combined With Warmed Intravenous Fluid on Core Temperature.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, In-Jung Jun, assistant professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-08-011-001
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Urologic Diseases
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warming group (Active Comparator): warming of the patient with whole body warming blanket in the OR during induction of anesthesia, prewarmed intravenous fluid during the operation.
  Interventions: Procedure: warming during induction of anesthesia; Procedure: Prewarmed intravenous fluid administration
- no warming group (No Intervention): There will be no whole body warming during induction.

INTERVENTIONS:
Procedure: warming during induction of anesthesia — Warming group patients are applied air-forced warming device (bair-hugger 43'C) with blanket (warm touch, COVIDIEN, full body blanket) during induction of anesthesia in the operation room.
  Arms: warming group
Procedure: Prewarmed intravenous fluid administration — Prewarmed intravenous fluid is connected.
  Arms: warming group

SUMMARY:
Hypothermia occurs frequently during general anesthesia. This study is to evaluate the efficacy of 10 minutes of prewarming during induction of general anesthesia during urologic surgery.

DETAILED DESCRIPTION:
Hypothermia is of continuous issue in patients undergoing general anesthesia. During urologic operation (transurethral resection of bladder and prostate), bladder irrigation worsens hypothermia. Hence, various methods including prewarming of the patient are used to maintain core temperature during operation.

Prewarming is found to be effective in maintaining core temperature perioperatively by increasing peripheral tissue heat content. However, applying more than 30 minutes of prewarming may be impractical as a clinical routine practice. Hence, developing simple and effective method to prevent hypothermia is expected.

Here, the investigators planned to examine the effect of active warming (10 minutes of warming during induction of general anesthesia and prewarmed intravenous fluid intraoperatively) on hypothermia in patients undergoing urologic operation under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing urologic surgery(transurethral resection of bladder, prostate)

Exclusion Criteria:

* moderate to severe cardiopulmonary, renal impairment
* previous thyroid disease
* any infection sign
* abnormal temperature prior to induction of general anesthesia (<36'C or >37.5'C)
* refusal to participate in the study
* unable to understand the study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
incidence of hypothermia at the end of the operation | approximately 1-2hours after induction (at the end of operation)
  number of patients with hypothermia (<36'C) using esophageal stethoscope will be recorded.

SECONDARY OUTCOMES:
change in temperature drop before and end of operation | on arrival at the OR upto 1-2hours after induction (at the end of the operation)
  change in core temperature will be observed
thermal comfort | upto 1hour after end of the operation (at discharge of postanesthesia care unit)
  thermal comfort scale ( 0= very cold, 5= fine, 10= very hot and uncomfortable) will be used.
incidence of shivering | upto 1 hour after end of the operation (on arrival at the postanesthesia care unit)
  4 point shivering scale (0=none, 1=core and neck shivering, 2= upper extremity 3= whole body) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: In-Jung Jun, MD, PhD, Principal Investigator — assistant professor
Locations (1):
- Sanggye paik hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No